CLINICAL TRIAL: NCT02266433
Title: A Double-blinded, Prospective, Randomized, Controlled Trial Comparing Dexamethasone Versus Ketorolac Injection for the Treatment of Local Inflammatory Hand and Upper Extremity Disorders
Brief Title: Dexamethasone Versus Ketorolac Injection for the Treatment of Local Inflammatory Hand and Upper Extremity Disorders
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: due to PI's change to private practice
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12-00878
Record Dates: First submitted 2014-09-18; First posted 2014-10-17 (Estimated); Results first posted 2020-11-02 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: DeQuervains Tenosynovitis; Lateral Epicondylitis; Tennis Elbow; Trigger Finger; Tenosynovitis; Inflammatory Disease
Keywords: DeQuervains Tenosynovitis; Lateral Epicondylitis; Tennis Elbow; Trigger Finger; Tenosynovitis; Inflammatory Disease; Dexamethasone; Ketorolac; Toradol
MeSH Terms: conditions — Tennis Elbow; Trigger Finger Disorder; Tenosynovitis | interventions — Ketorolac; Ketorolac Tromethamine; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm Receiving Dexamethasone Injection (Active Comparator): Dexamethasone will be administered as a peritendinous soft tissue injection of 1 mL of dexamethasone sodium phosphate (4mg/mL) and 0.5 mL (5mg) of 1% lidocaine.
  Dexamethasone will be administered as a peritendinous soft tissue injection of 1 mL of dexamethasone sodium phosphate (4mg/mL) and 0.5 mL (5mg) of 1% lidocaine
  Patients will be followed at the initial office visit, 4-weeks, 8-weeks, 12-weeks, and 6 months post injection to determine clinical response. A second injection can be given only once if the patient desires due to no clinical response at the 4 or 8-week follow-up.
  Interventions: Drug: Dexamethasone
- Arm Receiving Ketorolac Injection (Experimental): Ketorolac will be administered as a peritendinous soft tissue injection of 1 mL of ketorolac (30mg/mL) and 0.5 mL (5mg) of 1% lidocaine.
  Patients will be followed at the initial office visit, 4-weeks, 8-weeks, 12-weeks, and 6 months post injection to determine clinical response. A second injection can be given only once if the patient desires due to no clinical response at the 4 or 8-week follow-up.
  Interventions: Drug: Ketorolac

INTERVENTIONS:
Drug: Ketorolac — The proposed use of ketorolac in this study is outside of the FDA-approved indication and is the investigational agent in this study
  Ketorolac is a non-steroidal anti-inflammatory drug (NSAID). The approved indication for Ketorolac is for the short-term (≤5 days) management of moderately severe, acute pain that requires analgesia at the opioid level, usually in a postoperative setting. It is highly protein bound (99%) and is largely metabolized by the liver. In it's approved indication it is contraindicated for those with renal impairment, active peptic ulcer disease, pregnant or nursing females, individuals with NSAID hypersensitivity, or individuals at high risk for bleeding/clotting disorders.
  Other Names: Toradol
  Arms: Arm Receiving Ketorolac Injection
Drug: Dexamethasone — Dexamethasone is a synthetic corticosteroid and possesses glucocorticoid activity, and will be used within its labeled indication for this study: intra-articular or soft tissue injection for: synovitis of osteoarthritis, epicondylitis, acute nonspecific tenosynovitis. It is the active comparator in this study.
  In its approved indication there use limitations for immunocompromised individuals, pregnant females, persons with allergy to steroids, individuals with systemic fungal infections, and individuals with cerebral malaria. It is contra-indicated in systemic fungal infections, and hypersensitivity to any component of this product, including sulfites.
  Arms: Arm Receiving Dexamethasone Injection

SUMMARY:
The primary objective of this study is to compare local corticosteroid hand and elbow injections to placebo or ketorolac to determine if there is an equal or better reduction of symptoms for common orthopaedic upper extremity disorders including: De Quervain's tenosynovitis, trigger fingers, and tennis elbow (lateral epicondylitis). The investigators will enroll 780 subjects, divided equally into three arms for each disease process, and compare the efficacy of Ketorolac injections to Dexamethasone injections by measuring patient's functional status scores and pain scores at 0 weeks, 4 weeks, 8 weeks, 12 weeks, and 6 month followup periods, prospectively over time.

DETAILED DESCRIPTION:
Objectives: The primary objective of this study is to compare local corticosteroid hand and elbow injections to placebo or ketorolac to determine if there is an equal or better reduction of symptoms for common orthopaedic upper extremity disorders including: De Quervain's tenosynovitis, trigger fingers, and tennis elbow (lateral epicondylitis).

Number of Subjects: 780 total subjects:

• 260 subjects in each of the 3 treatment groups (De Quervain's tenosynovitis, trigger fingers and lateral epicondylitis) Diagnosis and Main Inclusion Criteria Subjects 18 years or older, with any of the following diagnoses: De Quervain's tenosynovitis, trigger fingers, or lateral epicondylitis

Study Product, Dose, Route, Regimen: Peritendinous soft tissue injection for De Quervain's tenosynovitis, trigger fingers and lateral epicondylitis:

• 1 mL of ketorolac (30mg/mL) and 0.5 mL (5mg) of 1% lidocaine Duration of administration Single administration, with a second injection permitted only once as subject desires due to no major clinical response at the 4 or 8-week follow-up.

Reference therapy: Standard of care peritendinous soft tissue injection for De Quervain's tenosynovitis, trigger fingers, and lateral epicondylitis:

• 1 mL of dexamethasone sodium phosphate (4mg/mL) and 0.5 mL (5mg) of 1% lidocaine

Statistical Methodology: The sample size as stated above was derived by a power analysis. A power analysis indicated that a total sample size of 200 patients randomized equally (1:1 randomization) to each treatment arm (i.e trigger finger, De Quervain's disease, and tennis elbow) without any blocking or stratification would provide 80% statistical power (alpha=.05, beta=0.20) to detect a 10% difference in mean Quick Disabilities of the Arm, Shoulder and Hand (quickDASH) scores between cohorts assuming a common standard deviation of 25% (effect size = 10/25 = 0.4). To account for an estimated 30% loss to follow-up, the investigators plan to enroll a total of 260 patients per treatment arm (i.e. trigger finger, De Quervain's disease, and tennis elbow). In total, there will be approximately 780 patients enrolled among all treatment arms.

1.1 Background Many orthopaedic hand disorders are comprised of different forms of tendonitis, tenosynovitis, and arthritis. The inflammatory processes of these disorders cause discomfort and functional impairment for patients. Decreasing the inflammatory response by use of splinting, physiotherapy, systemic anti-inflammatory agents, and local anti-inflammatory injections helps to alleviate some or all of the discomfort (2-4). Steroid injections are not entirely benign, and complications include tendon ruptures, subcutaneous fat atrophy, skin pigmentation changes, cartilage damage, and hyperglycemic responses in diabetics (9-11, 22-23). Studies have shown that ketorolac, a non-steroidal anti-inflammatory agent has a potent anti-inflammatory effect comparable to corticosteroids and a strong analgesic effect allowing for reduced opioid consumption postoperatively (7, 8). One could argue that the potent anti-inflammatory properties of ketorolac could be used to substitute for local corticosteroid injections in treating certain hand disorders. Given the side-effect profile for corticosteroids it may be beneficial to treat inflammatory disorders with local ketorolac injections. Nonsteroidal anti-inflammatory agents also have their known systemic adverse effects including gastric ulceration and intestinal bleeding as well as impairment of renal function. Most of these side effects are theoretically avoided with local tissue injections.

1.2 Study Drugs

Ketorolac:

The proposed use of ketorolac in this study is outside of the FDA-approved indication and is the investigational agent in this study

Ketorolac is a non-steroidal anti-inflammatory drug (NSAID). The approved indication for Ketorolac is for the short-term (≤5 days) management of moderately severe, acute pain that requires analgesia at the opioid level, usually in a postoperative setting. It is highly protein bound (99%) and is largely metabolized by the liver. In it's approved indication it is contraindicated for those with renal impairment, active peptic ulcer disease, pregnant or nursing females, individuals with NSAID hypersensitivity, or individuals at high risk for bleeding/clotting disorders.

Dexamethasone:

Dexamethasone is a synthetic corticosteroid and possesses glucocorticoid activity, and will be used within its labeled indication for this study: intra-articular or soft tissue injection for: synovitis of osteoarthritis, epicondylitis, acute nonspecific tenosynovitis. It is the active comparator in this study.

In its approved indication there use limitations for immunocompromised individuals, pregnant females, persons with allergy to steroids, individuals with systemic fungal infections, and individuals with cerebral malaria. It is contra-indicated in systemic fungal infections, and hypersensitivity to any component of this product, including sulfites.

Lidocaine:

Lidocaine is a local anesthetic of the amide type, and will be used within its labeled indication for this study: production of local or regional anesthesia by infiltration techniques such as percutaneous injection. It is to be given as concomitant therapy with both the investigational agent, ketorolac injection, and the standard of care therapy, dexamethasone injection.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be diagnosed with at least one of the following: trigger finger, de quervain's tenosynovitis, or tennis elbow (lateral epicondylitis)
* Patients age 18 years of age or older from all racial/ethnic types
* Patient who are both males and females
* Study participants will include any New York University employee or students as these individuals also can get hand and upper extremity pathology. It will be specifically reiterated to them that their academic status or grades, or employment will not be affected by their decision to participate in this study. Record of the participation cannot be linked to an academic record.

Exclusion Criteria:

* Patients had previous steroid injection at the site in question within 90 days of enrollment
* Patients with a history of gastric ulcers, renal impairment, allergy/hypersensitivity to non-steroidal anti-inflammatory (NSAID) or lidocaine derivative medications, immunocompromised patients (HIV/AIDs) and pregnant females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2012-08; Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Sapienza, MD, Principal Investigator — NYU Hospital for Joint Diseases; NYULMC
Locations (1):
- New York University School of Medicine, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients will be enrolled from the private office of orthopaedic hand surgeons (Dr. Paksima and Dr. Sapienza) and the resident hand clinic at NYU Hospital for Joint Diseases held at the 23rd street clinic.
Groups:
- Arm Receiving Dexamethasone Injection: Dexamethasone will be administered as a peritendinous soft tissue injection of 1 mL of dexamethasone sodium phosphate (4mg/mL) and 0.5 mL (5mg) of 1% lidocaine
  Patients will be followed at the initial office visit, 4-weeks, 8-weeks, 12-weeks, and 6 months post injection to determine clinical response. A second injection can be given only once if the patient desires due to no clinical response at the 4 or 8-week follow-up.
  Dexamethasone: Dexamethasone is a synthetic corticosteroid and possesses glucocorticoid activity, and will be used within its labeled indication for this study: intra-articular or soft tissue injection for: synovitis of osteoarthritis, epicondylitis, acute nonspecific tenosynovitis. It is the active comparator in this study.
- Arm Receiving Ketorolac Injection: Ketorolac will be administered as a peritendinous soft tissue injection of 1 mL of ketorolac (30mg/mL) and 0.5 mL (5mg) of 1% lidocaine.
  Patients will be followed at the initial office visit, 4-weeks, 8-weeks, 12-weeks, and 6 months post injection to determine clinical response. A second injection can be given only once if the patient desires due to no clinical response at the 4 or 8-week follow-up.
  Ketorolac: The proposed use of ketorolac in this study is outside of the FDA-approved indication and is the investigational agent in this study
Period: Overall Study
Arm/Group | Arm Receiving Dexamethasone Injection | Arm Receiving Ketorolac Injection
Started | 127 | 118
Completed | 68 | 65
Not Completed | 59 | 53
Not completed — Lost to Follow-up | 54 | 46
Not completed — Withdrawal by Subject | 5 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm Receiving Dexamethasone Injection | Arm Receiving Ketorolac Injection | Total
Number analyzed (Participants) | 127 | 118 | 245
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 93 | 88 | 181
  >=65 years | 34 | 30 | 64
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 83 | 167
  Male | 43 | 35 | 78
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Trigger Finger Treatment Group: EQVAS Score
Description: The EuroQol-visual analogue scale (EQ-VAS) is a vertical visual analogue scale that takes values between 100 (best imaginable health) and 0 (worst imaginable health), on which patients provide a global assessment of their health.
Time Frame: Baseline
Population: Certain participants withdrew or were lost to follow up, hence the lower overall number of participants analyzed and decrease in number of participants analyzed in certain time-points.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Arm Receiving Dexamethasone Injection: Dexamethasone will be administered as a peritendinous soft tissue injection of 1 mL of dexamethasone sodium phosphate (4mg/mL) and 0.5 mL (5mg) of 1% lidocaine.
  Dexamethasone will be administered as a peritendinous soft tissue injection of 1 mL of dexamethasone sodium phosphate (4mg/mL) and 0.5 mL (5mg) of 1% lidocaine
  Patients will be followed at the initial office visit, 4-weeks, 8-weeks, 12-weeks, and 6 months post injection to determine clinical response. A second injection can be given only once if the patient desires due to no clinical response at the 4 or 8-week follow-up.
  Dexamethasone: Dexamethasone is a synthetic corticosteroid and possesses glucocorticoid activity, and will be used within its labeled indication for this study: intra-articular or soft tissue injection for: synovitis of osteoarthritis, epicondylitis, acute nonspecific tenosynovitis. It is the active comparator in this study.
  In its approved indication there use limitations for immunocompromised
Arm/Group | Arm Receiving Dexamethasone Injection | Arm Receiving Ketorolac Injection
Number analyzed (Participants) | 86 | 88
score on a scale | 82.07 (16.25) | 82.30 (13.70)

2. Primary Outcome: Trigger Finger Treatment Group: EQVAS Score
Description: as for outcome 1
Time Frame: 4 weeks
Population: Certain participants withdrew or were lost to follow up, hence the decrease in number of participants analyzed in certain time-points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm Receiving Dexamethasone Injection | Arm Receiving Ketorolac Injection
Number analyzed (Participants) | 62 | 59
score on a scale | 82.79 (13.48) | 82.56 (13.77)

3. Primary Outcome: Trigger Finger Treatment Group: EQVAS Score
Description: as for outcome 1
Time Frame: 8 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm Receiving Dexamethasone Injection | Arm Receiving Ketorolac Injection
Number analyzed (Participants) | 30 | 31
score on a scale | 82.17 (13.31) | 81.61 (13.65)

4. Primary Outcome: Trigger Finger Treatment Group: EQVAS Score
Description: as for outcome 1
Time Frame: 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm Receiving Dexamethasone Injection | Arm Receiving Ketorolac Injection
Number analyzed (Participants) | 8 | 11
score on a scale | 93.50 (6.35) | 83.91 (7.82)

5. Primary Outcome: Trigger Finger Treatment Group: EQVAS Score
Description: as for outcome 1
Time Frame: 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm Receiving Dexamethasone Injection | Arm Receiving Ketorolac Injection
Number analyzed (Participants) | 8 | 14
score on a scale | 90.25 (8.48) | 75.79 (14.39)

6. Primary Outcome: Trigger Finger Treatment Group: QuickDASH Functional Scores
Description: The QuickDASH (Quick - Disabilities of the Arm, Shoulder and Hand) is an 11-question standardized survey used to assess a patient's overall functional status and is widely used in the practice of orthopaedic surgery as an analog measurement of a patient's functional ability. Scores range from 0-100, with 100 being the most poor functionality and 0 being the best. This will be assessed at every visit by having the patient fill out the survey and our team calculating the score at the end of the visit.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm Receiving Dexamethasone Injection | Arm Receiving Ketorolac Injection
Number analyzed (Participants) | 88 | 89
score on a scale | 28.56 (19.46) | 27.38 (20.71)

7. Primary Outcome: Trigger Finger Treatment Group: QuickDASH Functional Scores
Description: as for outcome 6
Time Frame: 4 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm Receiving Dexamethasone Injection | Arm Receiving Ketorolac Injection
Number analyzed (Participants) | 62 | 62
score on a scale | 28.73 (20.03) | 27.56 (18.75)

8. Primary Outcome: Trigger Finger Treatment Group: QuickDASH Functional Scores
Description: as for outcome 6
Time Frame: 8 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm Receiving Dexamethasone Injection | Arm Receiving Ketorolac Injection
Number analyzed (Participants) | 31 | 32
score on a scale | 23.61 (17.55) | 21.88 (15.43)

9. Primary Outcome: Trigger Finger Treatment Group: QuickDASH Functional Scores
Description: as for outcome 6
Time Frame: 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm Receiving Dexamethasone Injection | Arm Receiving Ketorolac Injection
Number analyzed (Participants) | 9 | 12
score on a scale | 15.65 (18.01) | 28.27 (28.29)

10. Primary Outcome: Trigger Finger Treatment Group: QuickDASH Functional Scores
Description: as for outcome 6
Time Frame: 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm Receiving Dexamethasone Injection | Arm Receiving Ketorolac Injection
Number analyzed (Participants) | 8 | 15
score on a scale | 21.04 (21.08) | 25.90 (22.35)

11. Primary Outcome: Trigger Finger Treatment Group: EuroQuol-5D (EQ-5D) Functional Score
Description: The EQ-5D (EuroQol five-dimension scale) is a 5 question survey with 3 potential responses per question, based on measuring a patient's overall quality of life. The responses are compiled into a numerical score ranging from 1 to -0.11, with 1 being the best and -0.11 being the worst in terms of quality of life. This survey will be administered to patients at each visit, along with the other surveys.
Time Frame: Baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm Receiving Dexamethasone Injection | Arm Receiving Ketorolac Injection
Number analyzed (Participants) | 88 | 89
score on a scale | 0.77 (0.13) | 0.78 (0.16)

12. Primary Outcome: Trigger Finger Treatment Group: EuroQuol-5D (EQ-5D) Functional Score
Description: as for outcome 11
Time Frame: 4 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm Receiving Dexamethasone Injection | Arm Receiving Ketorolac Injection
Number analyzed (Participants) | 62 | 62
score on a scale | 0.76 (0.16) | 0.78 (0.14)

13. Primary Outcome: Trigger Finger Treatment Group: EuroQuol-5D (EQ-5D) Functional Score
Description: as for outcome 11
Time Frame: 8 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm Receiving Dexamethasone Injection | Arm Receiving Ketorolac Injection
Number analyzed (Participants) | 31 | 32
score on a scale | 0.83 (0.10) | 0.82 (0.12)

14. Primary Outcome: Trigger Finger Treatment Group: EuroQuol-5D (EQ-5D) Functional Score
Description: as for outcome 11
Time Frame: 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm Receiving Dexamethasone Injection | Arm Receiving Ketorolac Injection
Number analyzed (Participants) | 9 | 12
score on a scale | 0.87 (0.10) | 0.81 (0.19)

15. Primary Outcome: Trigger Finger Treatment Group: EuroQuol-5D (EQ-5D) Functional Score
Description: as for outcome 11
Time Frame: 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm Receiving Dexamethasone Injection | Arm Receiving Ketorolac Injection
Number analyzed (Participants) | 8 | 15
score on a scale | 0.88 (0.10) | 0.77 (0.18)

16. Primary Outcome: Trigger Finger Treatment Group: VAS Pain Scores
Description: VAS (Visual Analogue Scale) pain score is a 0-10 numerical score assessing patient's subjective level of reported pain. The higher the score, the higher the pain level. This will be recorded from the patient's written response at every visit.
Time Frame: Baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm Receiving Dexamethasone Injection | Arm Receiving Ketorolac Injection
Number analyzed (Participants) | 88 | 94
score on a scale | 5.41 (2.65) | 4.79 (2.47)

17. Primary Outcome: Trigger Finger Treatment Group: VAS Pain Scores
Description: as for outcome 16
Time Frame: 4 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm Receiving Dexamethasone Injection | Arm Receiving Ketorolac Injection
Number analyzed (Participants) | 63 | 64
score on a scale | 4.20 (2.74) | 4.48 (2.63)

18. Primary Outcome: Trigger Finger Treatment Group: VAS Pain Scores
Description: as for outcome 16
Time Frame: 8 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm Receiving Dexamethasone Injection | Arm Receiving Ketorolac Injection
Number analyzed (Participants) | 30 | 31
score on a scale | 4.23 (2.72) | 3.53 (2.82)

19. Primary Outcome: Trigger Finger Treatment Group: VAS Pain Scores
Description: as for outcome 16
Time Frame: 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm Receiving Dexamethasone Injection | Arm Receiving Ketorolac Injection
Number analyzed (Participants) | 8 | 11
score on a scale | 2.25 (2.25) | 2.68 (2.63)

20. Primary Outcome: Trigger Finger Treatment Group: VAS Pain Scores
Description: as for outcome 16
Time Frame: 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm Receiving Dexamethasone Injection | Arm Receiving Ketorolac Injection
Number analyzed (Participants) | 8 | 15
score on a scale | 1.75 (3.49) | 3.07 (3.57)

21. Primary Outcome: Trigger Finger Treatment Group: Quinnell Grading Scores
Description: The Quinnell grading system monitors for trigger symptom improvement with a range of 0 (minumum) to 4 (maximum) with a higher number corresponding to worse symptoms: 0-normal movement of finger; 1-uneven movement; 2-active correctible locking of digit; 3-passively correctible locking; 4-fixed deformity.
Time Frame: Baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm Receiving Dexamethasone Injection | Arm Receiving Ketorolac Injection
Number analyzed (Participants) | 91 | 95
score on a scale | 1.67 (0.76) | 1.79 (0.86)

22. Primary Outcome: Trigger Finger Treatment Group: Quinnell Grading Scores
Description: as for outcome 21
Time Frame: 4 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm Receiving Dexamethasone Injection | Arm Receiving Ketorolac Injection
Number analyzed (Participants) | 65 | 60
score on a scale | 1.37 (0.89) | 1.55 (1.08)

23. Primary Outcome: Trigger Finger Treatment Group: Quinnell Grading Scores
Description: as for outcome 21
Time Frame: 8 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm Receiving Dexamethasone Injection | Arm Receiving Ketorolac Injection
Number analyzed (Participants) | 49 | 29
score on a scale | 1.63 (1.00) | 1.07 (0.87)

24. Primary Outcome: Trigger Finger Treatment Group: Quinnell Grading Scores
Description: as for outcome 21
Time Frame: 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm Receiving Dexamethasone Injection | Arm Receiving Ketorolac Injection
Number analyzed (Participants) | 8 | 9
score on a scale | 1.13 (0.99) | 1.22 (1.09)

25. Primary Outcome: Trigger Finger Treatment Group: Quinnell Grading Scores
Description: The Quinnell grading system monitors for trigger symptom improvement with a range of 0 (minimum) to 4 (maximum) with a higher number corresponding to worse symptoms: 0-normal movement of finger; 1-uneven movement; 2-active correctible locking of digit; 3-passively correctible locking; 4-fixed deformity.
Time Frame: 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm Receiving Dexamethasone Injection | Arm Receiving Ketorolac Injection
Number analyzed (Participants) | 7 | 12
score on a scale | 1.14 (1.46) | 0.67 (0.89)

26. Primary Outcome: DeQuervain's Treatment Group: EQ-VAS Score
Description: as for outcome 1
Time Frame: Baseline
Population: Certain participants were lost to follow up, hence the decrease in number of participants analyzed in weeks 4 and 8. There were not enough data points for 12-week and 6-month statistical analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm Receiving Dexamethasone Injection | Arm Receiving Ketorolac Injection
Number analyzed (Participants) | 31 | 15
score on a scale | 82.16 (13.91) | 79.45 (19.00)

27. Primary Outcome: DeQuervain's Treatment Group: EQ-VAS Score
Description: as for outcome 1
Time Frame: 4 weeks
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm Receiving Dexamethasone Injection | Arm Receiving Ketorolac Injection
Number analyzed (Participants) | 22 | 11
score on a scale | 26.19 (18.58) | 52.93 (14.55)

28. Primary Outcome: DeQuervain's Treatment Group: EQ-VAS Score
Description: as for outcome 1
Time Frame: 8 weeks
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm Receiving Dexamethasone Injection | Arm Receiving Ketorolac Injection
Number analyzed (Participants) | 10 | 3
score on a scale | 84.2 (12.68) | 87.33 (7.77)

29. Primary Outcome: De Quervain's Treatment Group: QuickDASH Scores
Description: as for outcome 6
Time Frame: Baseline
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm Receiving Dexamethasone Injection | Arm Receiving Ketorolac Injection
Number analyzed (Participants) | 31 | 17
score on a scale | 39.05 (19.51) | 47.40 (16.61)

30. Primary Outcome: De Quervain's Treatment Group: QuickDASH Scores
Description: as for outcome 6
Time Frame: 4 weeks
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm Receiving Dexamethasone Injection | Arm Receiving Ketorolac Injection
Number analyzed (Participants) | 21 | 11
score on a scale | 26.19 (18.58) | 52.93 (14.55)

31. Primary Outcome: De Quervain's Treatment Group: QuickDASH Scores
Description: as for outcome 6
Time Frame: 8 weeks
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm Receiving Dexamethasone Injection | Arm Receiving Ketorolac Injection
Number analyzed (Participants) | 11 | 3
score on a scale | 23.61 (16.18) | 68.34 (19.64)

32. Primary Outcome: DeQuervain's Treatment Group: EQ-5D Score
Description: as for outcome 11
Time Frame: Baseline
Population: Certain participants were lost to follow up, hence the decrease in number of participants analyzed in weeks 4 and 8.
  There was not enough data points for 12-week and 6-month statistical analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm Receiving Dexamethasone Injection | Arm Receiving Ketorolac Injection
Number analyzed (Participants) | 31 | 17
score on a scale | 0.75 (0.13) | 0.75 (0.15)

33. Primary Outcome: DeQuervain's Treatment Group: EQ-5D Score
Description: as for outcome 11
Time Frame: 4 weeks
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm Receiving Dexamethasone Injection | Arm Receiving Ketorolac Injection
Number analyzed (Participants) | 21 | 11
score on a scale | 0.83 (0.1) | 0.71 (0.18)

34. Primary Outcome: DeQuervain's Treatment Group: EQ-5D Score
Description: as for outcome 11
Time Frame: 8 weeks
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm Receiving Dexamethasone Injection | Arm Receiving Ketorolac Injection
Number analyzed (Participants) | 11 | 3
score on a scale | 0.85 (0.08) | 0.74 (0.13)

35. Primary Outcome: De Quervain's Treatment Group: VAS Pain Score
Description: VAS (Visual Analogue Scale) pain score is a 0-10 numerical score assessing patient's subjective level of reported pain. The higher the score, the higher and worse the pain level. This will be recorded from the patient's written response at every visit.
Time Frame: Baseline
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm Receiving Dexamethasone Injection | Arm Receiving Ketorolac Injection
Number analyzed (Participants) | 31 | 17
score on a scale | 7.03 (2.02) | 6.94 (1.99)

36. Primary Outcome: De Quervain's Treatment Group: VAS Pain Score
Description: as for outcome 35
Time Frame: 4 weeks
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm Receiving Dexamethasone Injection | Arm Receiving Ketorolac Injection
Number analyzed (Participants) | 23 | 10
score on a scale | 4.35 (2.28) | 5.35 (3.02)

37. Primary Outcome: De Quervain's Treatment Group: VAS Pain Score
Description: as for outcome 35
Time Frame: 8 weeks
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm Receiving Dexamethasone Injection | Arm Receiving Ketorolac Injection
Number analyzed (Participants) | 11 | 3
score on a scale | 3.05 (2.24) | 7.33 (0.58)

38. Primary Outcome: Lateral Epicondylitis Treatment Group: Participants With Pain (Positive Test) Over Lateral Epicondyle
Description: Clinician will examine the patient and palpate over the lateral epicondyle. Presence of pain is a positive test, recorded as 1. Absence of pain is a negative test, recorded as 0. This is done at every visit.
Time Frame: Baseline
Population: Certain participants withdrew or were lost to follow up, hence the lower overall number of participants analyzed and decrease in number of participants analyzed in certain time-points. Follow-up at 12-weeks and 6-months was not completed, as symptoms were resolved at week 8.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm Receiving Dexamethasone Injection | Arm Receiving Ketorolac Injection
Number analyzed (Participants) | 0 | 1
Participants |  | 1

39. Primary Outcome: Lateral Epicondylitis Treatment Group: Participants With Pain (Positive Test) in Lateral Epicondyle
Description: as for outcome 38
Time Frame: 4 weeks
Population: as for outcome 38
Measure: Count of Participants; unit: Participants
Arm/Group | Arm Receiving Dexamethasone Injection | Arm Receiving Ketorolac Injection
Number analyzed (Participants) | 0 | 1
Participants |  | 1

40. Primary Outcome: Lateral Epicondylitis Treatment Group: Participants With Pain (Positive Test) Over Lateral Epicondyle
Description: as for outcome 38
Time Frame: 8 weeks
Population: as for outcome 38
Measure: Count of Participants; unit: Participants
Arm/Group | Arm Receiving Dexamethasone Injection | Arm Receiving Ketorolac Injection
Number analyzed (Participants) | 0 | 1
Participants |  | 0

41. Primary Outcome: Lateral Epicondylitis Treatment Group: Participants With Pain (Positive Test) With Resisted Wrist Extension
Description: The clinician examines the patient and asks patient to extend wrist against resistance by the clinician. Production of pain is a positive test, recorded as 1. Absence of pain is a negative test, recorded as 0. This is done at every visit.
Time Frame: Baseline
Population: as for outcome 38
Measure: Count of Participants; unit: Participants
Arm/Group | Arm Receiving Dexamethasone Injection | Arm Receiving Ketorolac Injection
Number analyzed (Participants) | 0 | 1
Participants |  | 1

42. Primary Outcome: Lateral Epicondylitis Treatment Group: Participants With Pain (Positive Test) With Resisted Wrist Extension
Description: as for outcome 41
Time Frame: 4 weeks
Population: as for outcome 38
Measure: Count of Participants; unit: Participants
Arm/Group | Arm Receiving Dexamethasone Injection | Arm Receiving Ketorolac Injection
Number analyzed (Participants) | 0 | 1
Participants |  | 1

43. Primary Outcome: Lateral Epicondylitis Treatment Group: Participants With Pain (Positive Test) With Resisted Wrist Extension
Description: as for outcome 41
Time Frame: 8 weeks
Population: as for outcome 38
Measure: Count of Participants; unit: Participants
Arm/Group | Arm Receiving Dexamethasone Injection | Arm Receiving Ketorolac Injection
Number analyzed (Participants) | 0 | 1
Participants |  | 0

44. Primary Outcome: Lateral Epicondylitis Treatment Group: QuickDASH Functional Scores
Description: as for outcome 6
Time Frame: Baseline
Population: as for outcome 38
Measure: Number; unit: score on a scale
Arm/Group | Arm Receiving Dexamethasone Injection | Arm Receiving Ketorolac Injection
Number analyzed (Participants) | 0 | 1
score on a scale |  | 14

45. Primary Outcome: Lateral Epicondylitis Treatment Group: QuickDASH Functional Scores
Description: as for outcome 6
Time Frame: 4 weeks
Population: as for outcome 38
Measure: Number; unit: score on a scale
Arm/Group | Arm Receiving Dexamethasone Injection | Arm Receiving Ketorolac Injection
Number analyzed (Participants) | 0 | 1
score on a scale |  | 8

46. Primary Outcome: Lateral Epicondylitis Treatment Group: QuickDASH Functional Scores
Description: as for outcome 6
Time Frame: 8 weeks
Population: as for outcome 38
Measure: Number; unit: score on a scale
Arm/Group | Arm Receiving Dexamethasone Injection | Arm Receiving Ketorolac Injection
Number analyzed (Participants) | 0 | 1
score on a scale |  | 9

47. Primary Outcome: Lateral Epicondylitis Treatment Group: EQ-5D Scores
Description: as for outcome 11
Time Frame: Baseline
Population: as for outcome 38
Measure: Number; unit: score on a scale
Arm/Group | Arm Receiving Dexamethasone Injection | Arm Receiving Ketorolac Injection
Number analyzed (Participants) | 0 | 1
score on a scale |  | 0.83

48. Primary Outcome: Lateral Epicondylitis Treatment Group: EQ-5D Scores
Description: as for outcome 11
Time Frame: 4 weeks
Population: as for outcome 38
Measure: Number; unit: score on a scale
Arm/Group | Arm Receiving Dexamethasone Injection | Arm Receiving Ketorolac Injection
Number analyzed (Participants) | 0 | 1
score on a scale |  | 0.83

49. Primary Outcome: Lateral Epicondylitis Treatment Group: EQ-5D Scores
Description: as for outcome 11
Time Frame: 8 weeks
Population: as for outcome 38
Measure: Number; unit: score on a scale
Arm/Group | Arm Receiving Dexamethasone Injection | Arm Receiving Ketorolac Injection
Number analyzed (Participants) | 0 | 1
score on a scale |  | 1

50. Primary Outcome: Lateral Epicondylitis Treatment Group: VAS Pain Score
Description: as for outcome 35
Time Frame: Baseline
Population: as for outcome 38
Measure: Number; unit: score on a scale
Arm/Group | Arm Receiving Dexamethasone Injection | Arm Receiving Ketorolac Injection
Number analyzed (Participants) | 0 | 1
score on a scale |  | 6

51. Primary Outcome: Lateral Epicondylitis Treatment Group: VAS Pain Score
Description: as for outcome 35
Time Frame: 4 weeks
Population: as for outcome 38
Measure: Number; unit: score on a scale
Arm/Group | Arm Receiving Dexamethasone Injection | Arm Receiving Ketorolac Injection
Number analyzed (Participants) | 0 | 1
score on a scale |  | 4

52. Primary Outcome: Lateral Epicondylitis Treatment Group: VAS Pain Score
Description: as for outcome 35
Time Frame: 8 weeks
Population: as for outcome 38
Measure: Number; unit: score on a scale
Arm/Group | Arm Receiving Dexamethasone Injection | Arm Receiving Ketorolac Injection
Number analyzed (Participants) | 0 | 1
score on a scale |  | 3

53. Primary Outcome: Lateral Epicondylitis Treatment Group: EQ-VAS Score
Description: The EQ-VAS (EuroQol visual analog scale) is a vertical visual analogue scale that takes values between 100 (best imaginable health) and 0 (worst imaginable health), on which patients provide a global assessment of their health.
Time Frame: Baseline
Population: as for outcome 38
Measure: Number; unit: score on a scale
Arm/Group | Arm Receiving Dexamethasone Injection | Arm Receiving Ketorolac Injection
Number analyzed (Participants) | 0 | 1
score on a scale |  | 89

54. Primary Outcome: Lateral Epicondylitis Treatment Group: EQ-VAS Score
Description: as for outcome 53
Time Frame: 4 weeks
Population: as for outcome 38
Measure: Number; unit: score on a scale
Arm/Group | Arm Receiving Dexamethasone Injection | Arm Receiving Ketorolac Injection
Number analyzed (Participants) | 0 | 1
score on a scale |  | 85

55. Primary Outcome: Lateral Epicondylitis Treatment Group: EQ-VAS Score
Description: as for outcome 53
Time Frame: 8 weeks
Population: as for outcome 38
Measure: Number; unit: score on a scale
Arm/Group | Arm Receiving Dexamethasone Injection | Arm Receiving Ketorolac Injection
Number analyzed (Participants) | 0 | 1
score on a scale |  | 90

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Arm Receiving Dexamethasone Injection | Arm Receiving Ketorolac Injection
All-Cause Mortality (participants affected / at risk) | 0/127 | 0/118
Serious Adverse Events (participants affected / at risk) | 0/127 | 0/118
Other Adverse Events (participants affected / at risk) | 2/127 | 0/118
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm Receiving Dexamethasone Injection (N=127) | Arm Receiving Ketorolac Injection (N=118)
Skin discoloration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — minor skin discoloration at the site of injection
Redness and itching (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — developed redness and an itch in an adjacent finger several minutes after injection which resolved without further issue

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-31): https://cdn.clinicaltrials.gov/large-docs/33/NCT02266433/Prot_SAP_000.pdf